CLINICAL TRIAL: NCT05141344
Title: The Effect of Pre-emptive Oral Melatonin Versus Placebo on Postoperative Analgesia in Infants After Thoracotomy for Closed Cardiac Surgeries: A Randomized Controlled Study.
Brief Title: Effect of Oral Melatonin on Postoperative Analgesia After Thoracotomy in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, Associate professor of anesthesia ,surgical intensive care and pain management ,Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-101-2021
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Melatonin; Tablets

STUDY DESIGN:
Intervention Model Description: 50 patients will be divided into 2 equal groups
Who Masked: Participant, Care Provider, Investigator
Masking Description: The drugs will be given by an anesthetist who is not one of the observers to ensure blindness
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin group (Active Comparator): patients in this group will be premedicated One hour before the start of surgery by receiving 0.5mg/kg orally of melatonin (Melatonin 3 mg ), (the tablet will be dissolved in 5 ml of water, to be given by syringe 5ml) in the preoperative unit
  Interventions: Drug: Melatonin 3 MG Oral Tablet
- placebo group (Placebo Comparator): patients in group P (n =25 ) will receive a placebo( sugary tablets dissolved in 5ml of water by syringe 5 ml) one hour before the start of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 3 MG Oral Tablet — it will be given orally one hour preoperatively
  Arms: melatonin group
Drug: Placebo — sugar-coated tablets will be given one hour preoperatively
  Arms: placebo group

SUMMARY:
Thoracotomy pain is one of the severest pain that should be taken seriously, especially in children. (1) Inadequate postoperative pain management can compromise respiratory function, delay postoperative extubation, increase the cost and delay hospital discharge.

Opioids are the most commonly used analgesics to manage postoperative pain; however, they have many possible unfavorable side effects, such as nausea, vomiting, pruritus, and respiratory depression. (3) Melatonin is an endogenous indoleamine secreted by the pineal gland. It has several important physiological functions, including regulation of the circadian rhythms, modulation of season changes, antioxidant, anti-inflammatory, and anticonvulsant effects. (4)

DETAILED DESCRIPTION:
The analgesic effect of melatonin may be referred to as Gi-coupled melatonin receptors, to Gi-coupled opioid-l-receptors or gamma-aminobutyric acid (GABA) receptors with a consequential reduction in anxiety and pain. (5) Gitto and co-workers(6) hypothesized that melatonin may have beneficial effects as an analgesic effect in preterm newborns that are subject to painful procedures, such as endotracheal intubation and mechanical ventilation without detected side effects. Pro-inflammatory and anti-inflammatory cytokines related to pain were more in the common sedation and analgesia group than in melatonin-treated infants suggesting the use of melatonin as an adjunct analgesic therapy during procedural pain. (6) Therefore Melatonin may be a useful perioperative drug as it does not have any known undesirable serious adverse effects. (7)

To the best of investigators' knowledge, this is the first study investigating the effect of melatonin on postoperative pain scores after thoracotomy in infants.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology( ASA) I, II
* less than 18months.
* males and females.
* scheduled for thoracotomy for closed cardiac surgery.

Exclusion Criteria:

* airway abnormalities.
* heart failure.
* endocrine disorders.
* Patients with hypersensitivity to any drug.
* beta blockers, any analgesics recieved within 24 h before surgery, or any psychotropic drugs.
* hepatic, renal diseases neuromuscular disease,
* coagulopathy.
* a history of hyperthermia.
* infection at the site of the block.

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
total pethidine consumption 24 hours postoperatively. | 24 hours
  total dose of pethidine given to the patients over 24 hours postopertively

SECONDARY OUTCOMES:
the intraoperative fentanyl consumption | 2 hours
  total fentanyl doses in ug
Neonatal-Infant pain scale | 4 hours,6 hours,8 hours,12 hours,18 hours, 24 hours postoperatively
  0 no pain 0-3 mild pain 3-5 moderate pain 5-7 severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Amany Hassan Saleh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No